CLINICAL TRIAL: NCT00489268
Title: Micro-Layer Ablation of Barrett's Metaplasia- A Two-Phase, Multi-Center Trial - Extension of Follow-up to 5 Years
Acronym: AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Covidien, GI Solutions (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: David S. Utley, MD, BÂRRX Medical, Inc.
Organization: Medtronic - MITG (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-200
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Results first posted 2011-06-30 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Barrett Esophagus
Keywords: Barrett's Esophagus; Intestinal Metaplasia; Radiofrequency Ablation
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Phase I: 6 J/cm2 (Active Comparator): Subjects randomized to the energy density group of 6 J/cm2 through the HALO Ablation System.
  Interventions: Device: HALO Ablation System
- Phase I: 8 J/cm2 (Active Comparator): Subjects randomized to the energy density group of 8 J/cm2 through the HALO Ablation System.
  Interventions: Device: HALO Ablation System
- Phase I: 10 J/cm2 (Active Comparator): Subjects randomized to the energy density group of 10 J/cm2 through the HALO Ablation System.
  Interventions: Device: HALO Ablation System
- Phase I: 12 J/cm2 (Active Comparator): Subjects randomized to the energy density group of 12 J/cm2 through the HALO Ablation System.
  Interventions: Device: HALO Ablation System
- Phase II (Active Comparator): All Halo 360 treatments performed at 10 J/cm2 through the HALO Ablation System. All Halo 90 treatments performed at 12 J/cm2 through the HALO Ablation System.
  Interventions: Device: HALO Ablation System

INTERVENTIONS:
Device: HALO Ablation System — Phase I: 1-2 ablation visits; Phase II 1 to 12 months: 1-2 ablation visits; Phase II 12 to 30 months: 1-3 ablation visits Phase II 55-60 months: 0-1 ablation visit
  ******Phase I was a dosimetry study and Phase II used the preferred dose. The same intervention was used for each dose.
  Other Names: HALO360; HALO90

SUMMARY:
This study was conducted in 2 serial phases (dosimetry phase and effectiveness phase) to evaluate a balloon-based ablation device (HALO360) that delivers a pre-set amount of energy density (J/cm2) to barrett's tissue. The dosimetry phase evaluated the dose-response and the safety of delivering 6 to 12 J/cm2. The effectiveness phase used 10 J/cm2 delivered twice for all patients, followed by Esophagogastroduodenoscopy (EGD) with biopsies at 1, 3, 6, and 12 months. A second ablation procedure was performed if Barretts esophagus (BE) was present at 1 or 3 months. A complete response (CR) was defined as all biopsy specimens negative for Barrett's Esophagus at 12 months. The effectiveness phase of the present study was extended to a 2.5-year follow-up. This trial incorporated an opportunity for persistent BE to be treated with a focal ablation device (HALO90), achieving a CR in 98.4% of patients by the 2.5-year follow-up,the results of which were published . There is ample evidence that RadioFrequency Ablation (RFA) for Barrett's esophagus is effective and safe. Having additional follow-up (5 years) would add valuable information to the literature, thus aiding the physician in making patient management decisions about the appropriate follow-up interval after RFA.

DETAILED DESCRIPTION:
This study is intended to gather additional information regarding the performance of a bipolar balloon electrode device (HALO360) utilizing radiofrequency (RF) energy in the micro-layer ablation of Barrett's esophagus, a precancerous, metaplastic change in the esophageal lining. The device has received 510(k) clearance for specific indications, including the treatment of Barrett's esophagus.

This study is conducted in two phases and is intended to further evaluate the effect of micro-layer ablation of Barrett's metaplasia using a 510(k) cleared, bipolar, balloon electrode device. Phase I (n=30) is intended to provide additional information regarding the effects of three randomized treatment parameters (energy settings, Joules/cm2). Phase II (n=70) is intended to provide additional information regarding the effects of the optimal technique and energy density settings (Joules/cm2) determined from the 1-month endoscopy results of Phase I. Phase 2 primary endpoint was histological clearance of Barrett's (% patients). This trial incorporated an opportunity for persistent BE to be treated with a focal ablation device (HALO90), at the 2.5-year follow-up, achieving a CR in 98.4% of patients. Having additional follow-up (5 years) would add valuable information to the literature, thus aiding the physician in making patient management decisions about the appropriate follow-up interval after RFA. This study will allow collection of 5-year follow-up biopsies and, thereafter, offer RFA for any subject with persistent Barrett's.

Upon approval of the present amendment to the protocol (B-200-5 year extension) and the informed consent form (ICF) at each study site, subjects who participated in B-200-2.5 year extension and had a biopsy at 2.5 years after initial enrollment will be offered participation in this extension.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has documented histopathological diagnosis of Barrett's metaplasia (without dysplasia) as follows:

   * biopsies obtained less than 6 months prior to enrollment, and
   * biopsies obtained and reviewed at the investigator institution, and
   * biopsy protocol included at least 4 quadrant biopsies per 2 cm length of Barrett's metaplasia
2. Barrett metaplasia endoscopic length:

   Phase I : 2-3 cm Barrett's length (inclusive) Phase II: 2-6 cm Barrett's length (inclusive)
3. Age 18-75 years inclusive
4. Subject agrees to participate, fully understands content of informed consent form, and signs the informed consent form
5. Five year extension: All subjects who participated in B-200-2.5 year extension and had a biopsy at 2.5 years after initial enrollment (n=61) will be offered participation in this extension.

Exclusion Criteria:

1. Subjects is pregnant or planning a pregnancy
2. Esophageal stricture preventing passage of endoscope or catheter
3. Active esophagitis (Hetzel-Dent Grade III or IV) described as erosions or ulcerations encompassing more than 10% of distal esophagus
4. Barrett's metaplasia with dysplasia (any previous biopsy)
5. History or current diagnosis of malignancy of the esophagus
6. Prior radiation therapy to the esophagus, except head and neck region radiation therapy
7. Any previous ablative therapy within the esophagus (photodynamic therapy, multipolar electrical coagulation, argon plasma coagulation, laser treatment, or other)
8. Any previous endoscopic mucosal resection within the esophagus
9. Any previous esophageal surgery, except fundoplication
10. Esophageal varices
11. Subject has an implantable pacing device (examples; AICD, neurostimulator, cardiac pacemaker) and has not received clearance for enrollment in this study by specialist responsible for the pacing device
12. Participation in another clinical study in past 60 days
13. Subject suffers from unstable psychiatric disorder(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-11; Primary Completion 2007-02 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Fleischer, MD, Principal Investigator — Mayo Clinic
Locations (10):
- United States (9):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - UC Irvine Medical Center, Orange, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Gastrointestinal Associates, Knoxville, Tennessee
  - Tacoma Digestive Disease and Research Center, Seattle, Washington
- Ponce Gastroenterology Research, Ponce, Puerto Rico

REFERENCES:
- [Result] Sharma VK, Wang KK, Overholt BF, Lightdale CJ, Fennerty MB, Dean PJ, Pleskow DK, Chuttani R, Reymunde A, Santiago N, Chang KJ, Kimmey MB, Fleischer DE. Balloon-based, circumferential, endoscopic radiofrequency ablation of Barrett's esophagus: 1-year follow-up of 100 patients. Gastrointest Endosc. 2007 Feb;65(2):185-95. doi: 10.1016/j.gie.2006.09.033. PMID 17258973
- [Result] Fleischer DE, Overholt BF, Sharma VK, Reymunde A, Kimmey MB, Chuttani R, Chang KJ, Lightdale CJ, Santiago N, Pleskow DK, Dean PJ, Wang KK. Endoscopic ablation of Barrett's esophagus: a multicenter study with 2.5-year follow-up. Gastrointest Endosc. 2008 Nov;68(5):867-76. doi: 10.1016/j.gie.2008.03.008. Epub 2008 Jun 17. PMID 18561930
- [Result] Fleischer DE, Overholt BF, Sharma VK, Reymunde A, Kimmey MB, Chuttani R, Chang KJ, Muthasamy R, Lightdale CJ, Santiago N, Pleskow DK, Dean PJ, Wang KK. Endoscopic radiofrequency ablation for Barrett's esophagus: 5-year outcomes from a prospective multicenter trial. Endoscopy. 2010 Oct;42(10):781-9. doi: 10.1055/s-0030-1255779. Epub 2010 Sep 20. PMID 20857372

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: 6 J/cm^2: The HALO System is an option for eradication of the diseased epithelium of all three subclasses of Barrett's esophagus (non-dysplastic Intestinal Metaplasia (IM), Low-Grade Dysplasia (LGD) and High-Grade Dysplasia (HGD). The HALO Systems include the circumferential HALO360 Ablation System and the focal HALO90. The Ablation Catheter and Energy Generator work together to deliver energy to the tissue resulting in tissue coagulation. The HALO360 System is designed for longer segment diseased tissue (2 cm or greater) or as an initial treatment to ensure all Barrett's tissue or buried Barrett's glands are eliminated within the zone of intestinal metaplasia. The HALO90 System is designed for short segment Barrett's (2 cm or less) or for follow-up treatment for small Barrett's islands and tongues. In this group, subjects were randomized to the energy density group of 6 J/cm^2. They received a dose of 6 J/cm^2 during the course of this study.
- Phase I: 8 J/cm^2: In this group, subjects were randomized to the energy density group of 8 J/cm^2. They received a dose of 8 J/cm^2 during the course of this study.
- Phase I: 10 J/cm^2: In this group, subjects were randomized to the energy density group of 10 J/cm^2. They received a dose of 10 J/cm^2 during the course of this study.
- Phase I: 12 J/cm^2: In this group, subjects were randomized to the energy density group of 12 J/cm^2. They received a dose of 12 J/cm^2 during the course of this study.
- Phase II: In this group, subjects were randomized to the energy density group of 6 J/cm^2. All Halo 360 treatments performed at 10 J/cm^2; All Halo 90 treatments performed at 12 J/cm^2
Period: Overall Study
Arm/Group | Phase I: 6 J/cm^2 | Phase I: 8 J/cm^2 | Phase I: 10 J/cm^2 | Phase I: 12 J/cm^2 | Phase II
Started | 1 | 10 | 10 | 11 | 70
Completed | 1 | 10 | 9 | 11 | 50
Not Completed | 0 | 0 | 1 | 0 | 20

BASELINE CHARACTERISTICS:
Groups:
- Phase I: 6 J/cm^2: The HALO System is an option for eradication of the diseased epithelium of all three subclasses of Barrett's esophagus (non-dysplastic IM, LGD and HGD. The HALO Systems include the circumferential HALO360 Ablation System and the focal HALO90. The Ablation Catheter and Energy Generator work together to deliver energy to the tissue resulting in tissue coagulation. The HALO360 System is designed for longer segment diseased tissue (2 cm or greater) or as an initial treatment to ensure all Barrett's tissue or buried Barrett's glands are eliminated within the zone of intestinal metaplasia. The HALO90 System is designed for short segment Barrett's (2 cm or less) or for follow-up treatment for small Barrett's islands and tongues. In this group, subjects were randomized to the energy density group of 6 J/cm^2. They received a dose of 6 J/cm^2 during the course of this study.
- Phase I: 8 J/cm^2: The HALO System is an option for eradication of the diseased epithelium of all three subclasses of Barrett's esophagus (non-dysplastic IM, LGD and HGD. The HALO Systems include the circumferential HALO360 Ablation System and the focal HALO90. The Ablation Catheter and Energy Generator work together to deliver energy to the tissue resulting in tissue coagulation. The HALO360 System is designed for longer segment diseased tissue (2 cm or greater) or as an initial treatment to ensure all Barrett's tissue or buried Barrett's glands are eliminated within the zone of intestinal metaplasia. The HALO90 System is designed for short segment Barrett's (2 cm or less) or for follow-up treatment for small Barrett's islands and tongues. In this group, subjects were randomized to the energy density group of 8 J/cm^2. They received a dose of 8 J/cm^2 during the course of this study.
- Phase I: 10 J/cm^2: The HALO System is an option for eradication of the diseased epithelium of all three subclasses of Barrett's esophagus (non-dysplastic IM, LGD and HGD. The HALO Systems include the circumferential HALO360 Ablation System and the focal HALO90. The Ablation Catheter and Energy Generator work together to deliver energy to the tissue resulting in tissue coagulation. The HALO360 System is designed for longer segment diseased tissue (2 cm or greater) or as an initial treatment to ensure all Barrett's tissue or buried Barrett's glands are eliminated within the zone of intestinal metaplasia. The HALO90 System is designed for short segment Barrett's (2 cm or less) or for follow-up treatment for small Barrett's islands and tongues. In this group, subjects were randomized to the energy density group of 10 J/cm^2. They received a dose of 10 J/cm^2 during the course of this study.
- Phase I: 12 J/cm^2: The HALO System is an option for eradication of the diseased epithelium of all three subclasses of Barrett's esophagus (non-dysplastic IM, LGD and HGD. The HALO Systems include the circumferential HALO360 Ablation System and the focal HALO90. The Ablation Catheter and Energy Generator work together to deliver energy to the tissue resulting in tissue coagulation. The HALO360 System is designed for longer segment diseased tissue (2 cm or greater) or as an initial treatment to ensure all Barrett's tissue or buried Barrett's glands are eliminated within the zone of intestinal metaplasia. The HALO90 System is designed for short segment Barrett's (2 cm or less) or for follow-up treatment for small Barrett's islands and tongues. In this group, subjects were randomized to the energy density group of 12 J/cm^2. They received a dose of 12 J/cm^2 during the course of this study.
- Phase II: The HALO System is an option for eradication of the diseased epithelium of all three subclasses of Barrett's esophagus (non-dysplastic IM, LGD and HGD. The HALO Systems include the circumferential HALO360 Ablation System and the focal HALO90. The Ablation Catheter and Energy Generator work together to deliver energy to the tissue resulting in tissue coagulation. The HALO360 System is designed for longer segment diseased tissue (2 cm or greater) or as an initial treatment to ensure all Barrett's tissue or buried Barrett's glands are eliminated within the zone of intestinal metaplasia. The HALO90 System is designed for short segment Barrett's (2 cm or less) or for follow-up treatment for small Barrett's islands and tongues. In this group, subjects were randomized to the energy density group of 6 J/cm^2. All Halo 360 treatments performed at 10 J/cm^2; All Halo 90 treatments performed at 12 J/cm^2
- Total: Total of all reporting groups
Arm/Group | Phase I: 6 J/cm^2 | Phase I: 8 J/cm^2 | Phase I: 10 J/cm^2 | Phase I: 12 J/cm^2 | Phase II | Total
Number analyzed (Participants) | 1 | 10 | 10 | 11 | 70 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 10 | 8 | 7 | 54 | 80
  >=65 years | 0 | 0 | 2 | 4 | 16 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 1 | 18 | 21
  Male | 1 | 10 | 8 | 10 | 52 | 81
Region of Enrollment [Number; unit: participants]
  United States | 1 | 10 | 10 | 11 | 52 | 84
  Puerto Rico | 0 | 0 | 0 | 0 | 18 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Histological Clearance of Barrett's Metaplasia
Description: The primary study outcomes were defined as the percent of patients with complete histological response to intestinal metaplasia (IM) (CR-IM). CR-IM means complete eradication of IM (diseased epithelium). A patient was considered a Complete Responder (CR) if all biopsies (100%) were negative for intestinal metaplasia (CR-IM).
Time Frame: 5 year
Population: The analysis was done per protocol.
Measure: Number; unit: Percent of Participants
Arm/Group | Phase I: 6 J/cm^2 | Phase I: 8 J/cm^2 | Phase I: 10 J/cm^2 | Phase I: 12 J/cm^2 | Phase II
Number analyzed (Participants) | 1 | 10 | 10 | 11 | 70
Percent of Participants | 100 | 20 | 78 | 82 | 92

2. Secondary Outcome: Progression of Histological Grade
Description: Secondary outcomes of progression of histological grade was defined as proportion of participants who had progression of disease such as (i) prevalence of dysplasia; (ii) Kaplan-Meier CR-IM (Complete Response to Intestinal Metaplasia) survival analysis.
Time Frame: 5 year
Population: The analysis was done per protocol.
Measure: Number; unit: Percent of Participants
Arm/Group | Phase I: 6 J/cm^2 | Phase I: 8 J/cm^2 | Phase I: 10 J/cm^2 | Phase I: 12 J/cm^2 | Phase II
Number analyzed (Participants) | 1 | 10 | 10 | 11 | 70
Percent of Participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Adverse Events
Description: The secondary outcome adverse events was defined as any event that occurred during the course of the trial
Time Frame: 5 year
Population: The analysis was done per protocol.
Measure: Number; unit: Participants
Arm/Group | Phase I: 6 J/cm^2 | Phase I: 8 J/cm^2 | Phase I: 10 J/cm^2 | Phase I: 12 J/cm^2 | Phase II
Number analyzed (Participants) | 1 | 10 | 10 | 11 | 70
Participants | 0 | 0 | 7 | 0 | 28

4. Secondary Outcome: Percentage of Participants With Sub-squamous Intestinal Metaplasia
Description: The secondary outcome sub-squamous intestinal metaplasia was defined as prevalence of buried glandular mucosa in the esophagus.
Time Frame: 5 year
Population: The analysis was done per protocol.
Measure: Number; unit: Percent of Participants
Arm/Group | Phase I: 6 J/cm^2 | Phase I: 8 J/cm^2 | Phase I: 10 J/cm^2 | Phase I: 12 J/cm^2 | Phase II
Number analyzed (Participants) | 1 | 10 | 10 | 11 | 70
Percent of Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Phase I: 6 J/cm^2 | Phase I: 8 J/cm^2 | Phase I: 10 J/cm^2 | Phase I: 12 J/cm^2 | Phase II
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/10 | 0/10 | 0/11 | 0/70
Other Adverse Events (participants affected / at risk) | 0/1 | 0/10 | 0/10 | 0/11 | 0/70

LIMITATIONS AND CAVEATS:
Study had no concurrent control arm, biopsy forceps were not standardized for all cases, the original patient group comprised 70 patients, whereas 69 and 61 patients were available at 1 and 2.5 years, respectively, 60 eligible patients at 5 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No